CLINICAL TRIAL: NCT01510860
Title: Double-blind, Double-dummy, Randomised, Crossover, Multicentre Phase IV Clinical Study Comparing the Effect of Ursofalk 500 mg Tablets od Versus Ursofalk 250 mg Capsules od on Liver Enzymes in the Treatment of Primary Biliary Cirrhosis
Brief Title: Ursofalk Tablets (500 mg) Versus Ursofalk Capsules (250 mg) in the Treatment of Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: URT-15/PBC
Record Dates: First submitted 2012-01-12; First posted 2012-01-18 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2012-01

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ursodeoxycholic acid (UDCA)250 mg (Active Comparator): UDCA 250 mg capsule
  Interventions: Drug: UDCA (Ursodeoxycholic acid)
- Ursodeoxycholic acid (UDCA)500 mg (Experimental): UDCA 500 mg tablet
  Interventions: Drug: UDCA (Ursodeoxycholic acid)

INTERVENTIONS:
Drug: UDCA (Ursodeoxycholic acid) — 250 mg
  Arms: Ursodeoxycholic acid (UDCA)250 mg
Drug: UDCA (Ursodeoxycholic acid) — 500 mg
  Arms: Ursodeoxycholic acid (UDCA)500 mg

SUMMARY:
The purpose of this study is to compare the efficacy of Ursofalk 500 mg tablets versus Ursofalk 500 mg capsules in the treatment of Primary Biliary Cirrhosis (PBC).

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy
* Signed informed consent
* Histologically proven non-cirrhotic liver disease

Exclusion Criteria:

* histologically proven cirrhosis
* PBC stage II+IV
* Positive HIV serology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change of liver enzymes between baseline and the end of the treatment-period with Ursofalk 250 mg capsules and the end of treatment-period with Ursofalk 500 mg tablets. | Between baseline and week 24

SECONDARY OUTCOMES:
Quality of Life | Between baseline and week 24

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rust, MD, Principal Investigator — Klinikum Grosshadern Munich
Locations (1):
- Klinikum Grosshadern, Munich, Germany

REFERENCES:
- [Result] Hopf C, Grieshaber R, Hartmann H, Hinrichsen H, Eisold M, Cordes HJ, Greinwald R, Rust C. Therapeutic Equivalence of Ursodeoxycholic Acid Tablets and Ursodeoxycholic Acid Capsules for the Treatment of Primary Biliary Cirrhosis. Clin Pharmacol Drug Dev. 2013 Jul;2(3):231-6. doi: 10.1002/cpdd.24. Epub 2013 Apr 15. No abstract available. PMID 27121784